CLINICAL TRIAL: NCT03908008
Title: A Parallel, Active Drug Controlled, Double Blind, Randomized, Multi-center, Phase III Clinical Trial to Compare the Efficacy and Safety of MT10107 Versus BOTOX® in Treatment of Glabella Line
Brief Title: Efficacy and Safety Study of MT10107 in the Treatment of Glabella Line
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT_PRT_GL03
Record Dates: First submitted 2014-11-18; First posted 2019-04-09 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Glabellar Frown Lines
Keywords: Glabella line; Glabella lines; Botulinum Toxin
MeSH Terms: interventions — Botulinum Toxins, Type A; coretox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botox (Botulinum toxin type A) (Active Comparator): 20U of the investigational drug will be intramuscularly injected to 5 sites of the glabella line. Treatment will be conducted just once in visit 2.
  Interventions: Drug: Botox (Botulinum toxin type A); Drug: MT10107 (Botulinum toxin type A)
- MT10107 (Botulinum toxin type A) (Experimental): 20U of the investigational drug will be intramuscularly injected to 5 sites of the glabella line. Treatment will be conducted just once in visit 2.
  Interventions: Drug: Botox (Botulinum toxin type A); Drug: MT10107 (Botulinum toxin type A)

INTERVENTIONS:
Drug: Botox (Botulinum toxin type A) — 20U of the investigational drug will be intramuscularly injected to 5 sites of the glabella line. Treatment will be conducted just once in visit 2.
Drug: MT10107 (Botulinum toxin type A) — 20U of the investigational drug will be intramuscularly injected to 5 sites of the glabella line. Treatment will be conducted just once in visit 2.

SUMMARY:
This study design is a parallel, active drug controlled, double blind, randomized, multi-centered, phase III clinical trial to compare the efficacy and safety of MT10107 versus BOTOX® in treatment of glabella line.

DETAILED DESCRIPTION:
This study design is a parallel, active drug controlled, double blind, randomized, multi-centered, phase III clinical trial to compare the efficacy and safety of MT10107 versus BOTOX® in treatment of glabella line. Subjects who voluntarily signed the informed consent and are judged to be eligible for this study will be intramuscularly injected with the study drug or the comparator at a total of 20U (4U/0.1ml each) in five sites of the glabella line. Thereafter, follow-up visits will be made at 4 weeks, 10 weeks, 16 weeks and the efficacy and safety assessments will be conducted for a total of 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients attaining ≥grade 2(moderate) in the investigator's rating of the severity of glabella line at maximum frown
* Men and women aged between 20 and 65
* Patients who him/herself or him/her legal representatives voluntarily signed the informed consent
* Patients who can comply with the study procedures and visit schedule

Exclusion Criteria:

* Patients with general neuromuscular synaptic disorder(e.g. Myasthenia gravis, Lambert-Eaton syndrome, Amyotrophic lateral sclerosis)
* Patients who have bleeding tendency or taking anti-coagulant
* Patients suffering from acute diseases
* Patients who have been injected with botulinum toxin within past 3 months before the injection
* Patients with allergy or hypersensitivity to the investigational products or their components
* Patients who are pregnant or lactating or found to be pregnant through the urine or serum test or disagreed to avoid pregnancy during 16 weeks study period
* Patients who have been given any of the following drugs within previous 4 weeks at screening: Muscle relaxants, benzodiazepine, aminoglycoside antibiotics, other antibiotics, and anticholinergic drugs.
* Patients with the history of facial nerve paralysis or the symptoms of eyelid ptosis
* Patients with skin damage or infection at the injection site.
* Patients who scheduled a double eyelid operation during the clinical trial.
* Patients who have received or have a plan to receive other procedures, which may affect glabella and forehead lines within 6 months
* Patients whose glabella lines cannot be spread apart even with physical methods like using hands.
* Patients who are participating in other clinical trials or have participated in other clinical trials within 30 days of the screening date.
* Patients who are unable to communicate or follow the instructions
* Patients who are not eligible for this study at the discretion of the investigator

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Investigator's live assessment of glabella line improvement rate | 4 weeks after the injection
  Glabella line improvement rate determined by investigator's live assessment of glabella line severity at maximum frown at 4 weeks after the injection.

SECONDARY OUTCOMES:
Investigator's live assessment of glabella line improvement rate | 10, 16 weeks after the injection
  Glabella line improvement rate determined by investigator's live assessment of glabella line severity at maximum frown at 10, 16 weeks after the injection
Investigator's live assessment of glabella line improvement rate | 4, 10, 16 weeks after the injection
  Glabella line improvement rate determined by investigator's live assessment of glabella line severity at rest.
Investigator's photographic assessment of glabella line improvement rate at maximum frown | 4 weeks after the injection
  Glabella line improvement rate determined by investigator's photographic assessment of glabella line severity at maximum frown at 4 weeks after the injection.
Investigator's photographic assessment of glabella line improvement rate at rest | 4 weeks after the injection
  Glabella line improvement rate determined by investigator's photographic assessment of glabella line severity at rest.
Subject's satisfaction questionnaire to assess treatment efficacy | 4, 10, 16 weeks after the injection
  Subject's satisfaction questionnaire from score 1 to 7, with 7 being the most satisfied, to assess the glabella line improvement at 4, 10, 16 weeks after the injection.
Glabella line improvement rate of subject's assessment | 4, 10, 16 weeks after the injection
  Subject's assessment of glabella line improvement rate at 4, 10, 16 weeks after the injection.
The number of participants with adverse events determined by MedDra ver 17.0 for assessment of safety in IP | Through study completion, approximately 8 months
  The number of participants with adverse events determined by MedDra ver 17.0 for assessment of safety in IP from the study start date to the end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Huh Changhun, M.D., Study Chair — Seoul National University Bundang Hospital; Yangwon Lee, M.D., Principal Investigator — Konkuk University Hospital; Jonghee Lee, M.D., Principal Investigator — Samsung Medical Center